CLINICAL TRIAL: NCT05356013
Title: A Double-Blind, Placebo-Controlled Study of Caplyta in the Treatment of Borderline Personality Disorder
Brief Title: Caplyta in Borderline Personality Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB21-0974
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-05

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): All subjects who are randomized to Placebo will receive an identical placebo pill to the experimental drug starting the first week of the study. Subjects will be seen every two weeks for 8 weeks. After study conclusion (week 8), the dose will be discontinued.
  Interventions: Drug: Placebo
- Caplyta (Experimental): All subjects who are randomized to Caplyta will receive 42mg/day starting the first week of the study. Subjects will be seen every two weeks for 8 weeks. Dosage changes and reductions will not be permitted. After study conclusion (week 8), the dose will be discontinued.
  Interventions: Drug: Caplyta

INTERVENTIONS:
Drug: Caplyta — Atypical antipsychotic
  Other Names: lumateperone
  Arms: Caplyta
Drug: Placebo — Pill that contains no medicine.
  Other Names: no other names
  Arms: Placebo

SUMMARY:
The primary objective of the proposed study is to evaluate the safety and efficacy of Caplyta (lumateperone) in adults with borderline personality disorder (BPD). Sixty subjects with BPD will be randomized in a 1:1 fashion to either Caplyta (42mg/day) or matching placebo for 8 weeks of active treatment. The hypothesis to be tested is that Caplyta will result in greater rates of reduction in symptoms of BPD compared to placebo (improvement in symptoms will be indicated by lower scores on established outcome measures of BPD symptoms that have been used in prior studies).

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is a serious, difficult to treat, psychiatric disorder that causes significant emotional distress, as well as resulting in significant economic burden to health care systems. A variety of psychotherapies, particularly dialectical behavior therapy (DBT) and systems training for emotional predictability and problem solving (STEPPS), have shown benefit in reducing many of the core symptoms of BPD. Healthcare systems, however, often lack the funding and appropriate expertise to implement these treatments, and finding trained DBT or STEPPS therapists has been difficult for many people with BPD. While research on the use of medication is ongoing, no drug has yet been approved in the United States or elsewhere for the treatment of BPD. Antidepressants, anti-convulsants, and second generation antipsychotics have all been examined, but current medication options for BPD often provide only partial relief and may have pronounced side effects.

BPD is characterized by a pervasive pattern of severe psychopathological symptoms with instability of affect regulation, impulse control, and aggression. Dysfunctions in the serotoninergic, dopaminergic, and glutamatergic systems have been demonstrated in-and considered as possible causes for-symptoms associated with the disorder. Caplyta (lumateperone) therefore has distinctive properties that make it a promising option for patients with BPD. Caplyta is a mechanistically novel agent as it simultaneously modulates serotonin, dopamine, and glutamate, the key neurotransmitters implicated in BPD. Specifically, Caplyta acts as a potent serotonin 5-HT2A receptor antagonist, a dopamine D2 receptor pre-synaptic partial agonist and post-synaptic antagonist, a D1 receptor-dependent modulator of glutamate, and a serotonin reuptake inhibitor. In addition, because of low rates of side effects, Caplyta should be a well-tolerated and in fact desired medication approach to BPD.

The aim of the present study is to examine the efficacy and safety of Caplyta vs. placebo in adults with BPD, as indicated by a score of at least 9 on the Zanarini Rating Scale for Borderline Personality Disorder ("Zanarini scale"), a scale of illness severity, at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18-65;
2. Primary diagnosis of BPD
3. Zanarini scale score of at least 9 at baseline
4. Currently receiving for at least the last 2 months prior to study entry some form of weekly cognitive behavioral therapy
5. Ability to understand and sign the consent form.

Exclusion Criteria:

1. Unstable medical illness based on history or clinically significant abnormalities on baseline physical examination
2. Subjects with schizophrenia or bipolar I disorder
3. Subjects with an active substance use disorder
4. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
5. Subjects considered an immediate suicide risk based on the Columbia Suicide Severity rating Scale (C-SSRS) (www.cssrs.columbia.edu/docs)
6. Illegal substance use based on urine toxicology screening (excluding marijuana given the high rates of marijuana use in BPD and the lack of interaction with Caplyta).
7. Use of any new psychotropic medication started within the last 3 months prior to study initiation
8. Previous treatment with Caplyta
9. Cognitive impairment that interferes with the capacity to understand and self-administer medication or provide written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Zanarini Rating Scale for Borderline Personality Disorder | 8 Weeks
  A clinician-administered scale assessing Borderline Personality Scale severity

SECONDARY OUTCOMES:
Modified Overt Aggression Scale | 8 Weeks
  A clinician-administered behavior rating scale measuring four types of aggressive behavior that will be assessed at all 9 visits. The subsets range on a scale from 0-4 with 0 indicating no aggression present. This scale tracks changes in level of aggression over time. The total weighted sum of the sections of the scale is recorded. Higher total scores indicate higher aggression levels.
Young Mania Rating Scale | 8 Weeks
  A clinician-administered, 11 item scale that assesses manic symptoms at baseline and over time. Higher total scores indicate higher severity of manic symptoms. This scale is used to rate the severity of manic abnormality in the patient. Subsets of the scale range from 0-4 with 0 indicating no severity. This scale will be assessed at all visits.
Self-Report Version of Zanarini Scale | 8 Weeks
  A self-report scale assessing Borderline Personality severity that will be assessed at all 5 visits. This scale is assessing severity and change in BPD symptoms. Scoring is done by counting the number of yes's. A score of 8 or more is indicative of a diagnosis of borderline personality disorder.
Borderline Evaluation of Severity Over Time | 8 Weeks
  A self rated scale used to measure severity and change. The first 12 items of the scale are on a scale from 1-5, with 5 meaning that the item caused extreme distress, severe difficulties in relationships, and/or kept them from getting things done. The lowest rating (1) means it caused little or no problems. Items 13-15 (positive behaviors) are rated according to frequency. This scale will be assessed at all visits.
Barratt Impulsiveness Scale (BIS) | 8 Weeks
  A self-report assessment of impulsivity that will be assessed at baseline and Visit 5. All items are added to result in a total score. Higher total scores indicate higher impulsiveness.
Minnesota Impulsive Disorders Interview (MIDI) | 8 Weeks
  A clinical interview that screens for a variety of impulsive disorders, including buying disorder, kleptomania, trichotillomania, intermittent explosive disorder, pyromania, gambling disorder, compulsive sexual behavior, and binge eating disorder.
Symptom Checklist-90-Revised (SCL-90-R) | 8 Weeks
  An instrument that helps evaluate a broad range of psychological problems and symptoms of psychopathology. This will be assessed at baseline and visit 5.
Hamilton Depression Rating Scale | 8 Weeks
  A clinician-administered assessment of depression that will be assessed at all study visits. Higher total scores indicate higher levels of depression, while a score of 0 would indicate no depressive symptoms.
Hamilton Anxiety Rating Scale | 8 Weeks
  A clinician-administered assessment of anxiety that will be assessed at all study visits. Changes in scores from baseline to final visit will be assessed. Higher scores indicate higher levels of anxiety, with 0 being no symptoms of anxiety.
Quality of Life Inventory | 8 Weeks
  A self-report assessment of patient perceived quality of life that will be assessed at baseline and visit 5. Higher scores indicate a higher quality of life, whereas lower scores indicate a lower quality of life.
Sheehan Disability Scale (SDS) | 8 Weeks
  Subjects will complete the SDS at all visits. The change in scores from baseline to study completion will be assessed. The scale itself assesses the level of disability from borderline personality disorder (or target disorder) with higher scores indicating a more debilitating disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States